CLINICAL TRIAL: NCT02957617
Title: An Uncontrolled, Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability, and Maintenance of Effect of BIIB074 (Vixotrigine) in Subjects With Neuropathic Pain From Lumbosacral Radiculopathy
Brief Title: Extension Study to Evaluate the Long-Term Safety, Tolerability, and Maintenance of Effect of BIIB074
Acronym: RELAY-1 Extend
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The parent study did not meet its primary or secondary efficacy endpoints and therefore Sponsor decision to discontinue development in this indication.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1014802-204; 2015-004796-68 (EudraCT Number)
Record Dates: First submitted 2016-10-14; First posted 2016-11-08 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Neuropathic Pain From Lumbosacral Radiculopathy
Keywords: Neuropathic Pain From Lumbosacral Radiculopathy
MeSH Terms: interventions — vixotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIIB074 (Experimental): BIIB074 orally twice daily
  Interventions: Drug: BIIB074

INTERVENTIONS:
Drug: BIIB074 — Participants will receive an initial dose regimen of 350mg orally twice daily (BID), which may be reduced to 200mg based on tolerability for up to 12 months.
  Other Names: CNV1014802

SUMMARY:
The primary objective of the study is to evaluate the long-term safety and tolerability of BIIB074 in participants with neuropathic Pain From Lumbosacral Radiculopathy (PLSR). A secondary objective is to investigate the maintenance of effect during long-term treatment with BIIB074 in participants with neuropathic PLSR. For all efficacy assessments, baseline will be prior to randomization into Study 1014802-203. Another secondary objective is to evaluate the impact of treatment with BIIB074 on quality of life (QoL).

DETAILED DESCRIPTION:
This study was previously posted by Convergence Pharmaceuticals, Ltd., which has been acquired by Biogen. This is an extension study to 1014802-203.

ELIGIBILITY:
Key Inclusion Criteria:

* Has completed Study 1014802-203 for its complete duration.

Key Exclusion Criteria:

* Has met an exclusion criterion for the preceding double-blind Phase 2b study (Study 1014802-203).
* Had a protocol deviation regarding inclusion or exclusion criteria for the double-blind Phase 2b study (Study 1014802-203).
* Had a treatment-related AE or SAE that would pose an increased risk for continued treatment with BIIB074, or discontinued study treatment in the double-blind Phase 2b study (Study 1014802-203) due to an AE or SAE.
* Did not return for all study visits after discontinuing treatment in the double-blind phase of the Phase 2b study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants experiencing Adverse Events(AE) and Serious Adverse Events (SAEs) | Up to 395 Days
  Safety surveillance

SECONDARY OUTCOMES:
Change from Baseline to Week 52 in the weekly average of the daily neuropathic pain score on the Pain Intensity Numerical Rating Scale (PI-NRS) | Baseline to Week 52
  Participants will be asked every evening to rate their overall neuropathic pain for the last 24-hour period. PI-NRS is an 11-point pain intensity numerical rating scale (PI-NRS), where 0=no pain and 10=worst possible pain.
50% neuropathic pain reduction response | At Week 52
  Response is defined as a ≥50% reduction in the weekly average of the daily neuropathic pain score from Baseline to Week 52.
30% neuropathic pain reduction response | At Week 52
  Response is defined as a ≥30% reduction in the weekly average of the daily neuropathic pain score from Baseline to week 52.
Change from Baseline at each visit in the weekly average of the daily neuropathic pain score | Baseline through Week 52
  Participants will be asked every evening to rate their overall neuropathic pain for the last 24-hour period.
Change from Baseline to Week 52 in the weekly average of the daily pain score for low back pain | Baseline to Week 52
  Participants will be asked every evening to rate their overall low back pain for the last 24-hour period.
Number of Patient Global Impression of Change (PGIC) responder | At Week 52
  PGIC is a 7-point self-report scale depicting a participant's rating of overall improvement. Participants rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Change from Baseline to Week 52 on the Oswestry Disability Index (ODI) | Baseline to Week 52
  This is a 10-item questionnaire that evaluates how back (or leg) pain affects the ability to manage in everyday life. Each question is rated on a 5 point scale with higher scores indicating higher level of pain.
Change from Baseline to Week 52 in the weekly average of the daily sleep score as assessed by the Sleep Numerical Rating Scale (S-NRS) | Baseline to Week 52
  Participants will be asked every morning to rate on the 11-point S-NRS how leg pain interfered with their sleep quality where 0=no pain and 10=worst possible pain.
Change from Baseline to Week 52 in the Brief Pain Inventory (BPI)-Interference Index | Baseline to Week 52
  BPI Interference Index is an 11-point numeric rating scale (0 - no interference to 10 - interferes completely) to assess pain-related interference in 7 areas: general activity, mood, walking ability, normal work, including outside the home and housework, relations with other people, enjoyment of life and sleep.
Change from Baseline to Week 52 in the BPI - Pain Index | Baseline to Week 52
  BPI- Pain Index for pain intensity, is used to assess potential pain quality descriptors that may describe participants' pain on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
Change from Baseline to Week 52 on the EuroQoL 5-Dimension 5-Level Questionnaire (EQ-5D-5L) health index | Baseline to Week 52
  The EQ-5D-5L is a standardized instrument for use as a measure of health outcome. It is a health questionnaire that consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.
Change from Baseline to Week 52 in Short Form 36 Questionnaire (SF-36) | Baseline to Week 52
  SF-36 is a self-administered, generic health status questionnaire consisting of 36 questions that measure 8 health concepts: physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (37):
- Research Site, Klagenfurt, Austria
- Research Site, Leuven, Belgium
- Bulgaria (4):
  - Research Site, Blagoevgrad
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
- Czechia (8):
  - Research Site, Beroun
  - Research Site, Choceň
  - Research Site, Litoměřice
  - Research Site, Litomyšl
  - Research Site, Ostrava
  - Research Site, Prachatice
  - Research Site, Prague
  - Research Site, Zlín
- Research Site, Tartu, Estonia
- Research Site, Paris, France
- Research Site, Tbilisi, Georgia
- Research Site, Rome, Italy
- Latvia (2):
  - Research Site, Liepāja
  - Research Site, Riga
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
- Serbia (3):
  - Research Site 1, Belgrade
  - Research Site 2, Belgrade
  - Research Site, Belgrade
- Slovakia (5):
  - Research Site, Banská Bystrica
  - Research Site, Dubnica nad Váhom
  - Research Site, Krompachy
  - Research Site, Pruské
  - Research Site, Spišská Nová Ves
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid
- United Kingdom (3):
  - Research Site, Edinburgh
  - Research Site, Liverpool
  - Research Site, London